CLINICAL TRIAL: NCT05634993
Title: The Relationship Between Disability Level and Trunk Control in Individuals With Multiple Sclerosis
Brief Title: Disability Level and Trunk Control in Individuals With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Collaborators: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Melike Sumeyye Ozen, Research Assistant, Hacettepe University
Other Study IDs: 2022-42
Record Dates: First submitted 2022-11-11; First posted 2022-12-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; disability level; trunk control
MeSH Terms: conditions — Multiple Sclerosis | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MS Group
  Interventions: Other: Assessment

INTERVENTIONS:
Other: Assessment — Assessment of disability level and trunk control

SUMMARY:
Trunk control disorders are frequently encountered in individuals with MS. Trunk control is very important for safe and quality movement. Impairment of trunk control reduces the level of independence of individuals during activities of daily living. For this reason, it is extremely important to evaluate the trunk in the examination and treatment of individuals. When the literature was examined, it was seen that studies examining trunk control were insufficient. Therefore, our study was planned to investigate the relationship between disability level and trunk control in individuals with MS.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Having a definite diagnosis of MS
* Expanded Disability Status Scale (EDSS) score of 8.5 and below
* Not having an attack in the last 3 months

Exclusion Criteria:

* Having another musculoskeletal, cardiovascular, pulmonary, metabolic, or neurological disease severe enough to preclude participation in the study.
* Having severe vision and hearing problems
* The presence of severe cognitive impairment detected by the physician at a level that prevents the tests from being performed.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population of the study will consist of patients who applied to the Neurology Outpatient Clinic for outpatient treatment and were diagnosed with Multiple Sclerosis by a neurologist and volunteered to participate in the study.
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale | baseline
  It is used for the follow-up of neurological disability and disease stage in MS patients. A score of 0 on the scale indicates normal neurological status, while a score of 10 means death due to MS. The higher the score, the higher the disability level.
Trunk Impairment Scale | baseline
  This scale; It consists of 3 sub-headings: static sitting balance, dynamic sitting balance and coordination. The lowest score that can be obtained from the scale is 0, and the highest score is 23. The higher the score, the higher the trunk control.
"Sit-ups" test | baseline
  This test is used to evaluate the strength of the core stability muscles. Individuals are asked to flex the trunk while the knees are flexed in the supine position. The number of repetitions they can do for 30 seconds is recorded.
Modified "Push-ups" test | baseline
  This test is used to evaluate the strength of the core stability muscles. Individuals are asked to raise their body up by extending their elbows while in the prone position. The number of repetitions they can do for 30 seconds is recorded.
Lateral bridge test | baseline
  This test is used to evaluate the endurance of the core stability muscles. Individuals are asked to lift their bodies on their forearms and toes in the side-lying position and maintain this position. The time held in the position is recorded. The test is done separately for the right and left sides.
Modified "Biering-Sorensen" trunk extension test | baseline
  This test is used to evaluate the endurance of the core stability muscles. In the prone position, individuals are asked to hang their upper body over the edge of the bed and slightly extend them while their ankles are supported. The time held in the position is recorded.
Trunk flexion test | baseline
  This test is used to evaluate the endurance of the core stability muscles. Individuals are asked to stand with their torso at 60º with the floor, and their knees and hips at 90º. The time held in the position is recorded.
"Prone Bridge" test | baseline
  This test is used to evaluate the endurance of the core stability muscles.Individuals are asked to lift their torso up in the prone position while the elbows are flexed, carrying their body weight on their forearms and toes. The time held in the position is recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Melike Sumeyye Ozen, Bandırma, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No